CLINICAL TRIAL: NCT01236976
Title: SCIPA Full-On :Intensive Exercise Program After Spinal Cord Injury
Acronym: SCIPAFull-On
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Austin Health (Other Government); Hampstead Rehabilitation Centre Adelaide (Unknown); Shenton Park Rehabilitation Centre Perth (Unknown); Royal Rehabilitation Centre Sydney (Unknown); Prince of Wales Hospital, Sydney (Other Government); Burwood Hospital, Christchurch, New Zealand (Other)
Responsible Party: Principal Investigator, Mary Galea, Professor Mary Galea, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCIPA Full-On
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Participants in Group A will receive a triad of interventions comprising body weight supported treadmill training (BWSTT) using the Therastride Treadmill System, functional electrical stimulation (FES)-assisted cycling, and trunk and upper and lower limb exercise. These interventions will be provided at the spinal unit.
  Interventions: Device: Therastride Treadmill System; Device: FES-assisted cycling; Other: Trunk and upper and lower limb exercises
- Control Group (Other): Participants in Group B will receive an upper body strength and fitness program. This program may be provided at the spinal unit, or an appropriately equipped gymnasium as approved by the SCIPA Full-On Project Committee. It will be based on the Burn Rubber Burn (BRB) exercise program already established in Sydney. BRB is a circuit-based exercise program incorporating resistance and cardiovascular training. For this protocol, the circuit will comprise several stations using different pieces of equipment.
  Interventions: Other: Upper body strength and fitness program

INTERVENTIONS:
Device: Therastride Treadmill System — This device supports spinal cord injured patients to stand (suspended in a harness by an overhead pulley) on the specially designed treadmill for locomotor training. It is registered with the FDA (Regulation Number 890.5380).
  Arms: Intervention Group
Device: FES-assisted cycling — This intervention will be provided using a RT300 cycle (Restorative Therapies, Baltimore MD).
  Arms: Intervention Group
Other: Trunk and upper and lower limb exercises — This intervention will comprise assisted and/or resisted movements aimed at facilitating and strengthening voluntary muscle activity and improving movement quality.
  Arms: Intervention Group
Other: Upper body strength and fitness program — This intervention is a circuit-based exercise program incorporating resistance and cardiovascular training.
  Arms: Control Group

SUMMARY:
The study is a multi-centre, assessor-blind, randomised controlled phase III trial in patients with with complete or incomplete spinal cord injury between C6 and T12. A total of 188 participants will be randomised into two groups, the experimental group and the control group. The control group participants will receive an upper body strength and fitness program, conducted for 2-3 hours, three times per week for 12 weeks, while the experimental group participants will receive a comprehensive full body exercise program, conducted for 2-3 hours, three times per week for 12 weeks.

The main objective of this study is to determine if the experimental exercise program is more effective than the upper body strength and fitness program in promoting neurological improvement in participants with spinal cord injury.

Total study duration is 3.5 years, including a 24 month recruitment period, a 12-week treatment period followed by 6 month and 12 month (from baseline) follow up assessments.

Participants will be assessed by a blinded assessor (the assessor will not know which group the participants are in) using standard physiotherapy, neurophysiological, fitness and functional tests, psychological and quality of life questionnaires, as well as tests of immune function and bone structure.

DETAILED DESCRIPTION:
The study is a multi-centre, assessor-blind, randomised controlled phase III trial in patients with with complete or incomplete spinal cord injury between C6 and T12. A total of 188 participants will be randomised into two groups, the experimental group and the control group. The control group participants will receive an upper body strength and fitness program, conducted for 2-3 hours, three times per week for 12 weeks, while the experimental group articipants will receive a comprehensive full body exercise program, conducted for 2-3 hours, three times per week for 12 weeks.

The main objective of this study is to determine if the experimental exercise program is more effective than the upper body strength and fitness program in promoting neurological improvement in participants with spinal cord injury.

Total study duration is 3.5 years, including a 24 month recruitment period, a 12-week treatment period followed by 6 month and 12 month (from baseline) follow up assessments.

Participants will be assessed by a blinded assessor (the assessor will not know which group the participants are in) using standard physiotherapy, neurophysiological, fitness and functional tests, psychological and quality of life questionnaires, as well as tests of immune function and bone structure.

ELIGIBILITY:
Inclusion Criteria:

1. Have sustained a traumatic spinal cord injury a minimum of 6 months prior to consent and have completed their primary rehabilitation
2. Are 18 years or older and able to give informed consent
3. Have a complete or incomplete spinal cord injury between C6 and T12 (as per the International Standardised Neurological Assessment for SCI)
4. Are able and willing to attend an exercise program 3 times per week for 12 weeks
5. Are considered by their medical consultant to be fit to undertake the exercise program (documented approval by medical consultant required).

Exclusion Criteria:

1. Have brachial plexus, cauda equina, or peripheral nerve injury
2. Have had recent major trauma or surgery within the last 6 months
3. Have an existing pressure ulcer Stage 3 or 4 according to the National Pressure Ulcer Advisory Panel classification
4. Are post-menopausal at time of injury (females)
5. Have BMI at injury falling below lower threshold of healthy adult reference range
6. Have endocrinopathy or metabolic disorders of bone, such as Paget's disease, lytic or renal bone disease and senile osteoporosis
7. have medical history of exposure to medication(s) known to affect mineral ion or bone metabolism
8. Have chronic systemic diseases, e.g. Hep C, HIV-AIDs
9. Have significant impairment or disability, including physical, neurological or psychological impairments
10. Have a history of long bone fracture, or family history of fragility fracture
11. Have medical fragility, e.g. BMI falling below lower threshold of healthy adult reference range, or history of recurrent hospital readmissions.
12. Have extensive fixed contractures in upper or lower limbs
13. Have severe spasticity
14. Have uncontrolled neuropathic pain
15. Are likely to experience clinically significant autonomic dysreflexia and/or hypotension in response to electrical stimulation or prolonged upright posture
16. Are unable to attend the 6-month and 12 month follow-up assessments at their treating spinal unit
17. Have any contraindications to FES such as cardiac pacemaker, epilepsy, lower limb fracture or pregnancy
18. Have intracranial metal implants (for TMS only)
19. Have any other serious medical condition including malignancies, psychiatric, behavioural or drug-dependency problems, which are likely to influence the participant's ability to cooperate or in the opinion of the study investigator would prevent adherence to the Protocol.
20. Are participating in any other therapy (including alternative therapies) or taking medications (including herbal preparations) that are not considered to be standard care as per the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine the relative effectiveness of a comprehensive exercise program compared to a generic upper body strength and fitness training program on neurological improvement. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mary Galea, Principal Investigator — University of Melbourne; Prof Glen Davis, Principal Investigator — University of Sydney; Prof Sarah Dunlop, Principal Investigator — The University of Western Australia; Dr Andrew Nunn, Principal Investigator — Austin Health; Dr Tim Geraghty, Principal Investigator — Princess Alexandra Hospital Brisbane
Locations (6):
- Australia (5):
  - Spinal Unit, Prince of Wales Hospital, Randwick, New South Wales
  - Royal Rehabilitation Centre Sydney, Sydney, New South Wales
  - South Australian Spinal Cord Injury Service, Hampstead Rehabilitation Centre, Northfield, South Australia
  - Victorian Spinal Cord Injury Service, Royal Talbot Rehabilitation Centre, Kew, Victoria
  - Sir George Bebrook Spinal Injuries Centre, Royal Perth Hospital, Shenton Park, Western Australia
- Burwood Academy, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No
Aggregate data only. Individual participant data will not be provided as per the ethics approval.

REFERENCES:
- [Background] Galea MP, Dunlop SA, Davis GM, Nunn A, Geraghty T, Hsueh YS, Churilov L. Intensive exercise program after spinal cord injury ("Full-On"): study protocol for a randomized controlled trial. Trials. 2013 Sep 11;14:291. doi: 10.1186/1745-6215-14-291. PMID 24025260
- [Result] Galea MP, Dunlop SA, Geraghty T, Davis GM, Nunn A, Olenko L; SCIPA Switch-On Trial Collaborators<xref ref-type="fn" rid="fn1-1545968318771213" ptype="f1545968318771213" citart="citart1">*</xref>. SCIPA Full-On: A Randomized Controlled Trial Comparing Intensive Whole-Body Exercise and Upper Body Exercise After Spinal Cord Injury. Neurorehabil Neural Repair. 2018 Jun;32(6-7):557-567. doi: 10.1177/1545968318771213. Epub 2018 May 7. PMID 35545824